CLINICAL TRIAL: NCT06044519
Title: A Single Centre Randomized Control Trial of Donor Site Wound Dressing After Split Thickness Skin Grafting
Brief Title: A Single Center Trial of Donor Site Wound Dressings After Split Thickness Skin Grafting.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Approval/2022/943
Record Dates: First submitted 2023-09-04; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Donor Site Complication; Skin Graft Scar

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- alginate (Experimental)
  Interventions: Biological: different types of dressings
- film (Experimental)
  Interventions: Biological: different types of dressings
- guaze (Experimental)
  Interventions: Biological: different types of dressings
- hydrocolloid (Experimental)
  Interventions: Biological: different types of dressings
- hydrofiber (Experimental)
  Interventions: Biological: different types of dressings
- silicon (Experimental)
  Interventions: Biological: different types of dressings

INTERVENTIONS:
Biological: different types of dressings — different types of dressings were compared ti see the effectiveness for for STSG donor site wound

SUMMARY:
The goal of this clinical trial] is to compare different types of dressings used and there outcomes on STSG donor site wound. The main question[s] it aims to answer are:

* the effectiveness of different donor site dressings and their adverse outcomes
* the satisfaction of patients with the donor site dressing will be observed. Participants will randomly allocated different types of dressings for split thickness skin graft donor site wound which include alginate hydrocolloid hydrofiber silicon film guaze

ELIGIBILITY:
Inclusion Criteria:

* . Patients of aged 18 years and above of either gender underwent single donor-site wounds after split-skin grafting and surface area larger than 10 cm2 were included in the study

Exclusion Criteria:

* Patients on chemotherapy or corticosteroids were excluded from the study. Non-probability consecutive sampling was employed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
to asses the effective of dressings by measuring itching , pain and scarring | six month
  scaring by POSAS SCORE, pain and itcting by VISUAL ANALOGUE SCAORE.

SECONDARY OUTCOMES:
patient satisfaction for scar | six months
  likert scale
any complications | six months
  infection, hypergranulation, allergy

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Ruth KM Pfau civil hospital karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No